CLINICAL TRIAL: NCT04954456
Title: A Phase I Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of QLS31901 for Injection in Patients With Advanced Malignant Tumors
Brief Title: A Study of Bispecific Antibody QLS31901 in Patients With Advanced or Metastatic Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS31901-101
Record Dates: First submitted 2021-06-01; First posted 2021-07-08 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-06

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS31901 (Experimental): Part 1 (Dose escalation): QLS31901will be administered in sequential cohorts each receiving 1 of 6 doses of QLS31901 on day 1 of every 21-day cycle (3 weeks) via IV infusion. Dose escalation will continue until an MTD is reached.
  Part 2 (Dose Expansion): The PK parameters of QLS31901 will be tested at 2-3 doses determined during the dose-escalation phase in subjects with advanced malignant tumor cohorts.
  Interventions: Drug: QLS31901

INTERVENTIONS:
Drug: QLS31901 — QLS31901 is a bispecific antibody specifically targeting PD-L1 and TGF-β.In part 1,the QLS31901 will be administered in sequential cohorts on day 1 of every 21-day cycle (3 weeks) via IV infusion.In part 2,the QLS31901 will be administered in parallel cohorts(selected dose and dosing frequency ) on day 1 of every 2week or every 3week via IV infusion

SUMMARY:
This is a Phase 1, open label, non-randomised, dose-escalation single agent study with expansion cohorts for dose confirmation/safety and preliminary efficacy of QLS31901 in advanced or metastatic malignancies

DETAILED DESCRIPTION:
Study Design: This open label, multicenter, first in human study consists of 2 parts. Part 1 is a dose escalation to find the recommended dose for the expansion.

Part 2 is a dose expansion to confirm the dose of QLS31901 through further evaluation of safety, tolerability, Pk, preliminary antitumor activity, and functional target engagement.

The study includes three periods: Screening( up to 28 days prior to the first dose of study drug); Treatment(first dose of study drug with treatment cycles of 28 days); and Follow-up ( 30days 、60days and 90 days after the last dose) including survival follow-up checks every 3 months up to 12 months after the death of patient or the end of this clinical trial .

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years, male or female.
2. Eastern Cooperative Oncology Group (ECOG) score of 0-1.
3. Life expectancy ≥ 12 weeks.
4. At least one measurable lesion by imaging according to RECIST v1.1 evaluation criteria
5. Patients who failed standard treatment or were absent of standard treatment and have a pathologically confirmed advanced malignant tumor.
6. Sufficient organ function before the first dose of the investigational product

Exclusion Criteria:

1. Prior anti-cancer immunotherapy(Those who have received PD1 / PDL1 can be included in this study).
2. Known allergy to the investigational product or any excipient or severe anaphylaxis to other monoclonal antibodies.
3. Received any of the following treatments or drugs prior to the first dose of the study:
4. Symptomatic CNS metastasis, leptomeningeal metastases, or spinal cord compression due to metastasis before signing of the informed consent form.
5. Patients with uncontrollable severe exudation (thoracic cavity, pericardium, abdominal cavity);
6. Presence of active autoimmune disease or has a history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [patients whose condition can be controlled by thyroid hormone replacement therapy can be enrolled]; Subjects suffer from skin diseases that does not require systemic treatment, such as vitiligo, psoriasis, alopecia, type I diabetes, or childhood asthma that has completely alleviated and does not require any adult intervention can be enrolled. Asthmatic patients requiring bronchodilators for medical intervention cannot be enrolled);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 21days
  Safety and tolerability,as defined by the rate of treatment-related events as assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jifeng Feng, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China